CLINICAL TRIAL: NCT03419897
Title: A Phase 2, Open-label, Multicenter Study to Investigate the Efficacy, Safety, and Pharmacokinetics of the Anti-PD-1 Monoclonal Antibody BGB-A317 in Patients With Previously Treated Hepatocellular Unresectable Carcinoma
Brief Title: Study of BGB-A317 in Participants With Previously Treated Unresectable HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-208; 2017-003983-10 (EudraCT Number); CTR20171257 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Advanced liver cancer; RATIONALE-208
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental): 200 milligrams once every 3 weeks
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317

SUMMARY:
This study investigated the efficacy, safety, and pharmacokinetics of the anti-PD-1 monoclonal antibody BGB-A317 in participants with previously treated hepatocellular unresectable carcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed HCC
2. Participants with Barcelona Clinic Liver Cancer (BCLC) Stage C, or BCLC stage B not amenable to locoregional therapy or relapsed after locoregional therapy, and not amenable to a curative treatment approach
3. Has received at least 1 line of systemic therapy for unresectable HCC
4. Has at least 1 measurable lesion as defined per RECIST v1.1
5. Child-Pugh score A
6. Easter Cooperative Oncology Group (ECOG) Performance Status ≤ 1
7. Adequate organ function

Key Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC histology
2. Prior therapies targeting PD-1 or PD-L1
3. Has known brain or leptomeningeal metastasis
4. Tumor thrombus involving main trunk of portal vein or inferior vena cava
5. Loco-regional therapy to the liver within 4 weeks before enrollment
6. Medical history of interstitial lung disease, non-infectious pneumonitis or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, or acute lung diseases
7. Has received:

   1. Within 28 days or 5 half-lives (whichever is shorter) of the first study drug administration: any chemotherapy, immunotherapy (eg, interleukin, interferon, thymoxin) or any investigational therapies
   2. Within 14 days of the first study drug administration: sorafenib, regorafenib, or any Chinese herbal medicine or Chinese patent medicines used to control cancer
8. Active autoimmune diseases or history of autoimmune diseases that may relapse
9. Participant with any condition requiring systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication within 14 days before study drug administration

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (54):
- China (25):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Military Hospital of China, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- France (9):
  - Hopital Beaujon, Clichy
  - Hopital de La Croix Rousse, Lyon
  - Chu Montpellier Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital Larchet Chu Nice, Nice
  - Groupe Hospitalier Du Haut Leveque, Pessac
  - Chu de Poitiers Site de La Mileterie, Poitiers
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Kliniken Essen Mitte Evang Huyssens Stiftung, Essen
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Klinikum Johannes Gutenberg Universitaet Mainz, Mainz
- Italy (2):
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano
- Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw, Poland
- Spain (4):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Ico Lhospitalet Hospital Duran I Reynals, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid
- Taiwan (5):
  - E Da Hospital Kaohsiung, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - The Christie Hospital, Greater Manchester
  - Royal Free Hospital London Nhs Trust, London
  - Kings College, London
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ren Z, Ducreux M, Abou-Alfa GK, Merle P, Fang W, Edeline J, Li Z, Wu L, Assenat E, Hu S, Rimassa L, Zhang T, Blanc JF, Pan H, Ross P, Yen CJ, Tran A, Shao G, Bouattour M, Chen Y, Meyer T, Hou J, Tougeron D, Bai Y, Hou MM, Meng Z, Wu J, Li V, Chica-Duque S, Cheng AL. Tislelizumab in Patients with Previously Treated Advanced Hepatocellular Carcinoma (RATIONALE-208): A Multicenter, Non-Randomized, Open-Label, Phase 2 Trial. Liver Cancer. 2022 Oct 4;12(1):72-84. doi: 10.1159/000527175. eCollection 2023 Feb. PMID 36872927
- [Background] Serrano D, Podger L, Barnes G, Song J, Tang B. Psychometric validation of the EORTC QLQ-HCC18 in patients with previously treated unresectable hepatocellular carcinoma. Qual Life Res. 2022 Mar;31(3):937-950. doi: 10.1007/s11136-021-02992-1. Epub 2021 Sep 13. PMID 34518988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 73 study centers in Mainland China, Taiwan, Italy, Germany, France, Spain, Poland, and the United Kingdom.
Groups:
- Tislelizumab: Tislelizumab 200 milligrams (mg) administered intravenously once every 3 weeks until unacceptable toxicity, withdrawal of consent, or the time point at which the participant was no longer benefiting from therapy, as assessed by the investigator, whichever occurred first
Period: Overall Study
Arm/Group | Tislelizumab
Started | 249
Completed | 0
Not Completed | 249
Not completed — Death | 180
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Sponsor Decision | 61
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Tislelizumab: Tislelizumab 200 mg administered intravenously once every 3 weeks until unacceptable toxicity, withdrawal of consent, or the time point at which the participant was no longer benefiting from therapy, as assessed by the investigator, whichever occurred first
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 217
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 123
  White | 47
  Other | 1
  Not Reported | 78
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 129
    1 = Restricted Activity | 120

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assessed by Independent Review Committee (IRC)
Description: ORR is defined as the percentage of participants with complete response (CR) and partial response (PR) as the best overall response, as determined by an IRC using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR is defined as disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of first dose to primary analysis data cut-off date of 30-June-2021 (up to approximately 3 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants | 12.9 [8.96 to 17.66]
Statistical Analysis 1: Comparison: Tislelizumab; Tislelizumab compared with historical ORR rate of 7%; Test type: Superiority; p = 0.0001, Binomial exact test

2. Secondary Outcome: ORR Assessed by Investigator
Description: ORR is defined as the percentage of participants with CR and PR as the best overall response, as determined by investigator assessment using RECIST v1.1. CR is defined as disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants | 14.5 [10.34 to 19.45]

3. Secondary Outcome: Duration of Response (DOR) Assessed by IRC
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the IRC using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Months | NA [14.6 to NA] — Median DOR was not reached, and confidence interval data is not estimable due to insufficient number of participants with events

4. Secondary Outcome: DOR Event-Free Rate Assessed by IRC
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the IRC using RECIST v1.1. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for progression or death at 12 and 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months); Months 12 and 24 reported
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants
  12 Months | 76.9 [57.5 to 88.3]
  24 Months | 65.9 [45.7 to 80.1]

5. Secondary Outcome: DOR Assessed by Investigator
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the investigator using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Months | 21.4 [11.1 to NA] — Not estimable due to insufficient number of participants with events

6. Secondary Outcome: DOR Event-Free Rate Assessed by Investigator
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first, as assessed by the investigator using RECIST v1.1. The Kaplan-Meier method was used to estimate the percentage of participants who were event-free for progression or death at 12 and 24 months with 95% confidence intervals estimated using Greenwood's formula.
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months); Months 12 and 24 reported
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants
  12 Months | 68.1 [49.8 to 80.9]
  24 Months | 47.4 [30.1 to 62.8]

7. Secondary Outcome: Progression-free Survival (PFS) Assessed by IRC
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the IRC using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Months | 2.7 [1.4 to 2.8]

8. Secondary Outcome: PFS Assessed by Investigator
Description: PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the investigator using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Months | 2.8 [2.6 to 4.0]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first study drug administration to the date of death due to any cause
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Months | 13.2 [10.8 to 15.2]

10. Secondary Outcome: Disease Control Rate (DCR) Assessed by IRC
Description: DCR is defined as the percentage of participants whose best overall response is CR, PR, or stable disease (SD) as assessed by the IRC using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants | 53.0 [46.61 to 59.34]

11. Secondary Outcome: DCR Assessed by Investigator
Description: DCR is defined as the percentage of participants whose best overall response is CR, PR, or stable disease (SD) as assessed by the investigator using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants | 59.0 [52.65 to 65.20]

12. Secondary Outcome: Clinical Benefit Rate (CBR) Assessed by IRC
Description: CBR is defined as the percentage of participants who have CR, PR, or SD of ≥ 24 weeks in duration as assessed by the IRC using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants | 22.5 [17.46 to 28.19]

13. Secondary Outcome: CBR Assessed by Investigator
Description: CBR is defined as the percentage of participants who have CR, PR, or SD of ≥ 24 weeks in duration as assessed by the investigator using RECIST v1.1
Time Frame: From date of first dose to end of study (up to approximately 4 years and 3 months)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Percentage of participants | 30.9 [25.24 to 37.07]

14. Secondary Outcome: European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) Visual Analogue Score (VAS)
Description: Mean change from baseline in EQ-5D-5L VAS. The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 6 Day 1 and Cycle 12 Day 1 (each cycle is 21 days)
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug; "Overall number of participants analyzed" refers to number of participants evaluable for this outcome measure and "Number analyzed" refers to participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab
Number analyzed (Participants) | 202
Score on a scale
  Baseline | 75.2 (18.36)
  Change at Cycle 6: number analyzed (Participants) | 107
  Change at Cycle 6 | 2.4 (12.57)
  Change at Cycle 12: number analyzed (Participants) | 49
  Change at Cycle 12 | 4.7 (13.85)

15. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status
Description: Mean change from baseline in EORTC QLQ-C30 Global Health Status/Quality of Life score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of cancer patients. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 6 Day 1 and Cycle 12 Day 1 (each cycle is 21 days)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab
Number analyzed (Participants) | 238
Score on a scale
  Baseline | 71.8 (19.37)
  Change at Cycle 6: number analyzed (Participants) | 127
  Change at Cycle 6 | -0.1 (17.50)
  Change at Cycle 12: number analyzed (Participants) | 67
  Change at Cycle 12 | 1.1 (18.63)

16. Secondary Outcome: EORTC QLQ - Hepatocellular Carcinoma 18 Questions (HCC18): Index Scores
Description: Mean change from baseline in EORTC QLQ HCC18 Index Scores. The EORTC QLQ HCC18 is a specific questionnaire module that assesses quality of life of cancer patients related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 6 Day 1 and Cycle 12 Day 1 (each cycle is 21 days)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tislelizumab
Number analyzed (Participants) | 236
Score on a scale
  Baseline | 13.6 (11.33)
  Change at Cycle 6: number analyzed (Participants) | 129
  Change at Cycle 6 | 1.4 (11.77)
  Change at Cycle 12: number analyzed (Participants) | 60
  Change at Cycle 12 | 0.1 (8.27)

17. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), which includes laboratory tests, physical exams, electrocardiogram results and vital signs
Time Frame: From first dose up to 30 days after the last dose of study drug; up to approximately 4 years and 3 months
Population: Safety analysis set included all participants who received ≥ 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 249
Participants
  Participants with at least 1 TEAE | 236
  Participants with a serious TEAE | 94

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose of study drug (up to approximately 4 years and 3 months)
Description: Defined as an adverse event that had an onset date or worsening in severity from baseline (pretreatment) on or after the date of first dose of study drug up to 30 days after study drug discontinuation or initiation of new anticancer therapy.
Arm/Group | Tislelizumab
All-Cause Mortality (participants affected / at risk) | 180/249
Serious Adverse Events (participants affected / at risk) | 94/249
Other Adverse Events (participants affected / at risk) | 226/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tislelizumab (N=249)
Cardiac failure congestive (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Primary adrenal insufficiency (Endocrine disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 9
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemoperitoneum (Gastrointestinal disorders) | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Varices oesophageal (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 2
Death (General disorders) | 2
General physical health deterioration (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 2
Pyrexia (General disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Budd-Chiari syndrome (Hepatobiliary disorders) | 1
Hepatic artery aneurysm (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 7
Hepatic function abnormal (Hepatobiliary disorders) | 4
Hepatitis (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 2
COVID-19 (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Transaminases increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 2
Hepatic encephalopathy (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
VIth nerve paralysis (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Superior vena cava occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tislelizumab (N=249)
Anaemia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Hypothyroidism (Endocrine disorders) | 23
Abdominal distension (Gastrointestinal disorders) | 21
Abdominal pain (Gastrointestinal disorders) | 26
Abdominal pain upper (Gastrointestinal disorders) | 17
Ascites (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 30
Nausea (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 40
Fatigue (General disorders) | 28
Influenza like illness (General disorders) | 11
Oedema peripheral (General disorders) | 21
Pyrexia (General disorders) | 32
Nasopharyngitis (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 52
Aspartate aminotransferase increased (Investigations) | 66
Blood alkaline phosphatase increased (Investigations) | 21
Blood bilirubin increased (Investigations) | 48
Blood creatine phosphokinase MB increased (Investigations) | 14
Blood creatine phosphokinase increased (Investigations) | 10
Blood creatinine increased (Investigations) | 8
Blood lactate dehydrogenase increased (Investigations) | 11
Gamma-glutamyltransferase increased (Investigations) | 20
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 21
Total bile acids increased (Investigations) | 8
Weight decreased (Investigations) | 15
White blood cell count decreased (Investigations) | 17
Decreased appetite (Metabolism and nutrition disorders) | 43
Hyperglycaemia (Metabolism and nutrition disorders) | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18
Hypokalaemia (Metabolism and nutrition disorders) | 12
Hyponatraemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Back pain (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 17
Proteinuria (Renal and urinary disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 35
Rash (Skin and subcutaneous tissue disorders) | 24
Hypertension (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03419897/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03419897/SAP_001.pdf